CLINICAL TRIAL: NCT07279155
Title: A Study on the Bioequivalence of Bupivacaine Liposome Injection in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR-BBKY-BE-02
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Local Analgesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine liposome injection T preparation group (Experimental)
  Interventions: Drug: Bupivacaine Liposome Injection T preparation; Drug: Bupivacaine Liposome Injection R preparation
- Bupivacaine liposome injection R preparation group (Active Comparator)
  Interventions: Drug: Bupivacaine Liposome Injection T preparation; Drug: Bupivacaine Liposome Injection R preparation

INTERVENTIONS:
Drug: Bupivacaine Liposome Injection T preparation — Bupivacaine Liposome Injection T preparation
Drug: Bupivacaine Liposome Injection R preparation — Bupivacaine Liposome Injection R preparation
  Other Names: EXPAREL®

SUMMARY:
This study aims to investigate the pharmacokinetics of bupivacaine liposomal injection (test preparation) in healthy subjects. The manufactured liposomal bupivacaine injection (EXPAREL®) was used as the reference formulation to evaluate the human bioequivalence between the two formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between the ages of 18 and 45 years, inclusive;
2. At least 50.0 kg for male subjects, 45.0 kg for female subjects, with a Body Mass Index (BMI) between 19.0-26.0 kg/m2, inclusive (BMI = weight/height2);
3. Subjects (including male subjects) agree to adopt effective physical contraceptive measurements and not plan pregnancy, or sperm/ovum donation during the study till 90 days after the last administration. Pregnancy tests of female subjects must be negative before and during the study and female subjects were not lactating. (see Section 14.2 for details);
4. Subjects who could understand the nature, significance, potential benefits, inconvenience, and potential risks of the study, understand the procedures and methods, be willing to complete the trial strictly following the protocol, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Subjects with specific allergic diseases (asthma, urticaria, eczema, etc.) or allergic constitution (such as allergy to two or more drugs, food or pollen), or allergy to excipients and bupivacaine;
2. Subjects with history of serious diseases including but not limited to circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic disorders;
3. Abnormalities at the injection site (including skin diseases, open wounds, inflammation, scars, tattoos, etc.), which may affect the drug absorption;
4. Subjects who had undergone major trauma surgery within 6 months before the screening, or planned a surgery during the study;
5. Using any drugs that inhibit or induce the metabolism of drugs in liver within 30 days before the study (such as: inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors: SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones and antihistamines);
6. Use of any medication within 14 days prior to dosing (including vitamin products and herbal medicines);
7. Subjects who have taken any clinical investigational products or participated in the clinical research of medical devices within 3 months before the trial, or plan to participate in other clinical trials during the study;
8. Blood donation or massive loss (≥ 200 ml, excluding blood loss during menstrual period), received blood transfusion or blood products within 3 months before the trial;
9. Subjects who take more than 5 cigarettes per day on average within 3 months prior to the study or do not agree to prohibit smoking during the study;
10. Drinking frequently within 6 months before the trial, meaning 14 units of alcohol per week（1 unit = 360 mL beer or 45 mL of 40% spirits, or 150 mL wine), or disagree with the prohibition of alcohol during the study;
11. Subjects who were positive in drug abuse or had a history of drug abuse or use of illegal drugs within the past five years;
12. Clinical significance in vital signs, physical examination, ECG and clinical laboratory tests (chemistry, hematology, urinalysis, coagulation function);
13. Positive results in any one of Hepatitis B virus surface antigen, hepatitis C virus antibody, HIV antibody or syphilis serum reagin test;
14. Difficulty in venous blood collection or unable to tolerate venipuncture or abdominal subcutaneous injection;
15. Consumption of any special diet within 48 hours prior to dosing (including grapefruit, chocolate, xanthine rich food / beverage) and / or excessive consumption of tea, coffee, grapefruit juice, caffeinated beverage (more than 8 cups per day, 200 mL per cup) for the past three months;
16. Breath test for alcohol > 0.0 mg /mL;
17. Unable to complete the study due to personal reasons or other factors considered by the investigator as unsuitable to participate in the study (such as inability to understand the study requirements, poor compliance, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax). | From 0 hour predose up to 240 hours postdose.
  Blood samples will be collected.
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t). | From 0 hour predose up to 240 hours postdose.
  Blood samples will be collected.
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞). | From 0 hour predose up to 240 hours postdose.
  Blood samples will be collected.

SECONDARY OUTCOMES:
Observed time to reach Cmax (Tmax). | From 0 hour predose up to 240 hours postdose.
  Blood samples will be collected.
Adverse events (AEs). | From 0 hour predose up to 35 days postdose.

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided